CLINICAL TRIAL: NCT00044863
Title: A Phase II Multicenter Study of Erbitux (Cetuximab) in Patients With Metastatic Colorectal Carcinoma
Brief Title: Study of Erbitux (Cetuximab) in Patients With Metastatic Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP02-0144
Record Dates: First submitted 2002-09-05; First posted 2002-09-09 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Colorectal Neoplasms; Metastases, Neoplasm
Keywords: EGFr; Metastatic Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients with metastatic EGFR-positive colorectal carcinoma
  Interventions: Biological: Erbitux (Cetuximab)

INTERVENTIONS:
Biological: Erbitux (Cetuximab) — 400 mg/m2 initial dose, 250 mg/m2 weekly

SUMMARY:
This is a phase II, multicenter, target enrollment of 250 evaluable patients, open-label study of cetuximab in patients with refractory, metastatic colorectal carcinoma. Based on prior studies, we predict that 70 to 75% of patients will be EGFR-positive. Patients must have documented failure after receiving either at least two chemotherapy regimens for metastatic disease or adjuvant therapy plus one chemotherapy regimen for metastatic disease provided that the patient progressed within 6 months of completing adjuvant therapy. Prior chemotherapy must have included irinotecan, oxaliplatin, and a fluoropyrimidine.

Patients will receive an initial dose of cetuximab, 400 mg/m2, intravenously (i.v.) over 120 minutes, followed by weekly treatment with cetuximab, 250 mg/m2 i.v. over 60 minutes. Patients who experience unacceptable toxicity or who have progressive disease will not receive further cetuximab therapy.

Patients will be evaluated for a tumor response at a minimum of every 6 weeks while on cetuximab therapy. Patients with stable disease or a partial or complete response may continue to receive weekly cetuximab therapy, unless they are dose-delayed or discontinued because of toxicity. Patients who have a partial or complete response must have a confirmatory tumor assessment no less than 4 weeks after the initial evaluation demonstrating a response.

In addition, there is a pharmacokinetic companion protocol which will determine the trough and peak levels of cetuximab in 25 patients enrolled in the study at four to eight centers. A pharmacologic serum sample for the determination of levels of cetuximab will be obtained prior to the initial, fourth and sixth cetuximab infusions and 1 hour following the completion of the initial, fourth and sixth cetuximab infusions in the first course; and prior to and 1 hour post the completion of the first cetuximab infusion of each subsequent course of therapy. A course of therapy is defined as six weekly infusions of cetuximab monotherapy. ImClone will perform the pharmacokinetic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent.
* Histologically- or pathologically- confirmed metastatic colorectal carcinoma;
* Documented progressive disease after receiving either:

  1. at least two chemotherapy regimens for metastatic disease or
  2. adjuvant therapy plus one chemotherapy regimen for metastatic disease provided that the patient progressed within 6 months of completing adjuvant therapy. Progressive disease will be defined as progression while on treatment or within 3 months after receiving the last dose of therapy in a given regimen;
* Prior chemotherapy must have included irinotecan, oxaliplatin, and a fluoropyrimidine;
* Measurable disease as defined in Section 3.3.2;
* Immunohistochemical evidence of EGFr expression. Patients will be considered eligible if their tumors demonstrate any EGFr staining, regardless of the intensity, the cellular localization of the staining, or the percentage of cell staining. Patients who do not have tumor tissue available for EGFr testing will undergo biopsy of accessible tumor;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1 at study entry;
* Adequate recovery from recent surgery, chemotherapy, and radiation therapy. At least 4 weeks must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent, or prior radiation therapy;
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center;
* Men and woman age 18 years or older

Source documentation of the prior treatment (e.g., hospital/clinic records, radiographic reports) must be available to ImClone for review.

Exclusion Criteria:

Sex and Reproductive Status Exceptions

* Women of child bearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to cetuximab administration.
* Sexually active fertile men not using effective birth control.

Medical History and Concurrent Diseases

* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent;
* A serious uncontrolled medical disorder that would impair the ability of the patient to receive protocol therapy;
* A history of uncontrolled angina, arrhythmias, congestive heart failure, or left ventricular ejection fraction (LVEF) below the institutional range of normal on a baseline multiple gated acquisition (MUGA) scan or echocardiogram (ECHO);
* Known brain metastases;
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for greater than or equal to 5 years will be allowed to enter the trial;

Physical and Laboratory Test Findings

* Inadequate hematologic function defined by an absolute neutrophil count (ANC) <1,500/mm3, a platelet count <100,000/mm3, and a hemoglobin level <9 g/dL.
* Inadequate hepatic function, defined by a total bilirubin level greater than or equal to 1.5 times the upper limit of normal (ULN) and aspartate transaminase (AST) and alanine transaminase (ALT) levels greater than or equal to 5 times the ULN.
* Inadequate renal function defined by a serum creatinine level >1.5 times the ULN.

Prohibited Therapies and/or Medications

* A history of cetuximab or other therapy that targeted the EGF receptor;
* A history of prior anti-cancer murine monoclonal antibody therapy;
* Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2002-08; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Determine the response rate of cetuximab in patients with EGFR-positive, metastatic carcinoma | every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (1):
- ImClone Investigational Site, Saint Charles, Missouri, United States

REFERENCES:
- [Result] Zhang W, Gordon M, Schultheis AM, Yang DY, Nagashima F, Azuma M, Chang HM, Borucka E, Lurje G, Sherrod AE, Iqbal S, Groshen S, Lenz HJ. FCGR2A and FCGR3A polymorphisms associated with clinical outcome of epidermal growth factor receptor expressing metastatic colorectal cancer patients treated with single-agent cetuximab. J Clin Oncol. 2007 Aug 20;25(24):3712-8. doi: 10.1200/JCO.2006.08.8021. PMID 17704420
- [Result] Lenz HJ, Van Cutsem E, Khambata-Ford S, Mayer RJ, Gold P, Stella P, Mirtsching B, Cohn AL, Pippas AW, Azarnia N, Tsuchihashi Z, Mauro DJ, Rowinsky EK. Multicenter phase II and translational study of cetuximab in metastatic colorectal carcinoma refractory to irinotecan, oxaliplatin, and fluoropyrimidines. J Clin Oncol. 2006 Oct 20;24(30):4914-21. doi: 10.1200/JCO.2006.06.7595. PMID 17050875
- [Result] Vallbohmer D, Zhang W, Gordon M, Yang DY, Yun J, Press OA, Rhodes KE, Sherrod AE, Iqbal S, Danenberg KD, Groshen S, Lenz HJ. Molecular determinants of cetuximab efficacy. J Clin Oncol. 2005 May 20;23(15):3536-44. doi: 10.1200/JCO.2005.09.100. PMID 15908664